CLINICAL TRIAL: NCT06564168
Title: Nutritional Status of Critically Ill Diabetic Patients With Type 2 Diabetes Mellitus.
Brief Title: Nutritional Status of Critically Ill Diabetic Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Salwa Ahmed Mohammed Ali, Physician, Assiut University
Other Study IDs: Nutrition in Diabetes Mellitus
Record Dates: First submitted 2024-08-16; First posted 2024-08-21 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Nutrition; Critical Illness; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Critical Illness; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Crtitically ill Patients with diabetes mellitus type 2.
- Controls: All critically ill patients not Diabetes mellitus type 2.

SUMMARY:
1. To investigate the nutritional status of patients with type 2 diabetes mellitus in the intensive care unit.
2. To detect the impact of nutritional status on outcome (mortality, length of hospital stay,duration of mechanical ventilation, and need for renal replacement therapy)

DETAILED DESCRIPTION:
Nutrition support in the Intensive Care Unit is very important since it has a significant impact on recovery from illness and overall outcome. Patients in the intensive care unit have a higher risk of malnutrition than patients undergoing general admission to hospitals . In critically ill patients, malnutrition may result in impaired immunological function, impaired ventilatory drive, and weakened respiratory muscles, leading to prolonged ventilatory dependence and increased infectious morbidity and mortality.

An appropriate nutritional support is indispensable to critically ill patients, who are almost at the hyper-metabolic state of their clinical condition such as trauma, sepsis, and major surgery. These critical conditions result in a disproportional release of cytokine and stress hormones that alter energy and protein metabolism and eventually lead to malnourishment.

A recent systematic review revealed the strikingly high prevalence of malnutrition in intensive care unit patients (ranged from 38% to 78%), which is associated with the patients' increased morbidity, mortality, and hospital-related cost.The increased dependency on mechanical ventilation, length of hospital stay, intensive care unit readmission, persistence of infection, and risk of hospital mortality associated with undernutrition, make it an important dilemma in the care of Intensive Care unit patients.

Diabetes is a chronic disease that occurs either when the pancreas does not produce enough insulin or when the body cannot effectively use the insulin it produces. Insulin is a hormone that regulates blood glucose.( and associated with serious complications, demand for multimodal treatment, and significant economic burden With the development of complications and hospital lengths of stay, life expectancy is worsened with diabetes, and nutritional status is generally correlated with these total outcomes.

In this research,investigators will evaluate the nutritional state in critically ill diabetic patients with type 2 diabetes mellitus, and detect the impact of poor nutritional status on out comes regarding mortality, length of hospital stay , length of mechanical ventilation, and need for renal replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

Age above 18 years. Diabetic type ll. Admitted for more than 48 hours.

Exclusion Criteria:

Type 1 Diabetes Mellitus. Age under 18 years Readmission in intensive care unit. Adimssion for less than 48 hours

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who are admitted to the intensive care unit will be enrolled and divided into two groups. Group 1: includes all candidates with type 2 diabetes and meet the inclusion criteria and group 2: the control group includes patients without diabetes.
  All patients after informed consent will be subjected to:
  A: History. B: Examination. C: laboratory data: urea and creatinine, liver function test, and complete blood count.
  D: Nutritional status assessment scores:
  1. Nutritional risk score (NRS)-2002.
  2. Nutrition Risk in Critically ill (NUTRIC) score.
Sampling Method: Non-Probability Sample
Enrollment: 430 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Correlation between Diabetes Mellitus and malnutrition in critically ill patients | through study completion, an average of 1 year]
  By using non invasive methods to find a correlation between Diabetes mellitus and malnutrition in critically ill patients by history and examination and scores of nutrition
Outcome of patients with Diabetes Mellitus admitted in intensive care unit | through study completion, an average of 1 year]
  As Diabetic patiants are more suspectible to face malnutrition in intensive care unit so non invasive methods as history, examination, score to improve outcome and decrease morbidity and mortality.

REFERENCES:
- [Background] Sioson MS, Martindale R, Abayadeera A, Abouchaleh N, Aditianingsih D, Bhurayanontachai R, Chiou WC, Higashibeppu N, Mat Nor MB, Osland E, Palo JE, Ramakrishnan N, Shalabi M, Tam LN, Ern Tan JJ. Nutrition therapy for critically ill patients across the Asia-Pacific and Middle East regions: A consensus statement. Clin Nutr ESPEN. 2018 Apr;24:156-164. doi: 10.1016/j.clnesp.2017.11.008. Epub 2018 Jan 3. PMID 29576355
- [Background] Hoffer LJ, Bistrian BR. Nutrition in critical illness: a current conundrum. F1000Res. 2016 Oct 18;5:2531. doi: 10.12688/f1000research.9278.1. eCollection 2016. PMID 27803805
- [Background] Wray CJ, Mammen JM, Hasselgren PO. Catabolic response to stress and potential benefits of nutrition support. Nutrition. 2002 Nov-Dec;18(11-12):971-7. doi: 10.1016/s0899-9007(02)00985-1. PMID 12431720
- [Background] Lew CCH, Yandell R, Fraser RJL, Chua AP, Chong MFF, Miller M. Association Between Malnutrition and Clinical Outcomes in the Intensive Care Unit: A Systematic Review [Formula: see text]. JPEN J Parenter Enteral Nutr. 2017 Jul;41(5):744-758. doi: 10.1177/0148607115625638. Epub 2016 Feb 2. PMID 26838530
- [Background] Mogensen KM, Horkan CM, Purtle SW, Moromizato T, Rawn JD, Robinson MK, Christopher KB. Malnutrition, Critical Illness Survivors, and Postdischarge Outcomes: A Cohort Study. JPEN J Parenter Enteral Nutr. 2018 Mar;42(3):557-565. doi: 10.1177/0148607117709766. Epub 2017 Dec 18. PMID 28521598
- [Background] American Diabetes Association. Economic costs of diabetes in the U.S. In 2007. Diabetes Care. 2008 Mar;31(3):596-615. doi: 10.2337/dc08-9017. PMID 18308683
- See also: Global Burden of Disease Collaborative Network. Global Burden of Disease Study 2019. Results. Institute for Health Metrics and Evaluation. 2020 — https://vizhub.healthdata.org/gbd-results/).